## Informed Consent Form

Infections in migrants: the importance of malaria and other parasites

2020-10-27

## Consent form

## Informed consent for participation in the study: Infections in migrants - the importance of malaria and other parasites

To be signed before inclusion in the study.

I hereby certify that I have been informed about the study and given written information.

I am willing to participate in the study and I have understood that my participation is voluntary and that I can end my participation at any point without explanation.

## I approve

that the blood samples collected from me will be stored in Stockholm Medical Biobank according to the biobanking regulations

that the blood samples collected from me will be used in analyses described in the study information

that I at any point can withdraw my consent and that I can demand that my blood samples will be destroyed or anonymized

that the blood samples can be used in future biomedical research that is not described only after ethical approval from the Regional Committee for Research Ethics

that my personal data are registered in accordance with the General Data Protection Regulation (GDPR).

| Date | <br> |
|------------------------------------|------|
| Name | <br> |
| Personal identification number | |
| Signature | <br> |
| For children younger than 15 years | |
| Guardians name | <br> |
| Guardian's signature | |

This document is made in 2 originals, one is to be kept by the volunteering study participant and the other by the researcher.